CLINICAL TRIAL: NCT06258252
Title: Effect of Metabolic Dysfunction in Branched-chain Amino Acids on Cardiac Function in Patients With Sepsis: an Observational Study
Brief Title: Effect of Metabolic Dysfunction in Branched-chain Amino Acids on Cardiac Function in Patients With Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 20240201
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who are diagnosed as sepsis, with type 2 diabetes.: 1. myocardial injury-related biomarkers: troponin T and B natriuretic peptide levels; 2. cardiac structure-related indicators: the size of the left and right ventricle, left ventricular ejection fraction, etc.3. septic cardiomyopathy incidence: Troponin T>0.01ng/ml is the standard for the diagnosis of septic cardiomyopathy.
  Interventions: Other: Effect of BCAAs metabolic dysfunction on cardiac function in sepsis
- Patients who are diagnosed as sepsis, without type 2 diabetes.: 1. myocardial injury-related biomarkers: troponin T and B natriuretic peptide levels; 2. cardiac structure-related indicators: the size of the left and right ventricle, left ventricular ejection fraction, etc.3. septic cardiomyopathy incidence: Troponin T>0.01ng/ml is the standard for the diagnosis of septic cardiomyopathy.
  Interventions: Other: Effect of BCAAs metabolic dysfunction on cardiac function in sepsis

INTERVENTIONS:
Other: Effect of BCAAs metabolic dysfunction on cardiac function in sepsis — Effect of BCAAs metabolic dysfunction on cardiac function in sepsis

SUMMARY:
The current project was designed to examine the effects of BCAA metabolic dysfunction on cardiac function in septic patients.

DETAILED DESCRIPTION:
Patients with sepsis and with/without type 2 diabetes will be included. Patients prospectively collected the following indicators in the intensive care unit: 1. myocardial injury-related biomarkers: troponin T and B natriuretic peptide levels; 2. cardiac structure-related indicators: the size of the left and right ventricle, left ventricular ejection fraction, etc.3. septic cardiomyopathy incidence: Troponin T>0.01ng/ml is the standard for the diagnosis of septic cardiomyopathy. Additionally, the investigators will collect the peripheral blood at preoperative, day 1, day 3, and day 5 after surgery. Peripheral blood plasma and PBMCs were separated by differential centrifugation: the concentration of BCAAs in serum and PBMCs; the expression of PBMCs BCAAs metabolic enzymes BCAT 1, BCKDH, and PP 2 Cm by WB; and the levels of AST, ALT, LDH, CK, and CK-MB

ELIGIBILITY:
Inclusion Criteria:

- patients diagnosed with sepsis with or without type 2 diabetes

Exclusion Criteria:

- patients with immunodeficient diseases patients who accept glucocorticoid or immunosuppressant patients with an age younger than 18 years patients who cannot provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of Sepsis induced cardiomyopathy | up to 7 days post-ICU admission, or at hospital discharge, whichever comes first
  Diagnostic criteria for Sepsis induced cardiomyopathy, TroponinT > 0.01 ng/ml

SECONDARY OUTCOMES:
Plasma levels of TroponinT | up to 7 days post-ICU admission, or at hospital discharge, whichever comes first
  If multiple measurements is available during the first 7 days, the mean measurement will be used for analysis.
Plasma levels of type B natriuretic peptide | up to 7 days post-ICU admission, or at hospital discharge, whichever comes first
  If multiple measurements is available during the first 7 days, the mean measurement will be used for analysis.
ejection fraction | up to 7 days post-ICU admission, or at hospital discharge, whichever comes first
  If multiple measurements is available during the first 7 day, the mean measurement will be used for analysis.
Left ventricular and right ventricular size | up to 7 days post-ICU admission, or at hospital discharge, whichever comes first
  If multiple measurements is available during the first 7 day, the mean measurement will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fengmin Luo, PhD, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No